CLINICAL TRIAL: NCT00608088
Title: Support for Low-Income Breastfeeding: Cost and Outcomes
Brief Title: Evaluation of a Community Health Nurse/Peer Counselor Program to Help Low-Income Women Breastfeed Longer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Gayle G. Page RN, DNSc, FAAN, Johns Hopkins University School of Nursing
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: FWA 0006088; NIH/NINR - R01 RN007675
Record Dates: First submitted 2008-01-24; First posted 2008-02-06 (Estimated); Last update posted 2008-02-06 (Estimated); Status verified 2008-01

CONDITIONS: Breastfeeding Rates
Keywords: Breast feeding; breastfeeding; randomized clinical trial; poverty
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Usual Care
  Interventions: Behavioral: Usual Care
- 2 (Active Comparator): Health Nurse/Peer Councelor Intervention
  Interventions: Behavioral: Community Health Nurse/Peer Councelor Team

INTERVENTIONS:
Behavioral: Usual Care — The usual care group will received standard care from the Johns Hopkins Hospital lactation consultant and nurses, which may have included a visit in the hospital by the lactation consultant if mothers delivered Monday through Friday. The lactation consultant was also available by request. A "warm-line" was also standard. This was a telephone line that was connected to an answering machine; the lactation consultant checked this line once daily (Monday through Friday) and returned calls.
  Arms: 1
Behavioral: Community Health Nurse/Peer Councelor Team — Visits by a community health nurse/peer counselor team during the first six postpartum months. Based on prior research and experience, the team was developed to provide culturally relevant support and health-care education to low-income mothers, who were a high percentage of African American women. The goals of this team were to 1) increase the duration of breastfeeding while emphasizing ways to decrease fatigue, and decrease breast discomfort; 2) strengthen maternal competence with breastfeeding and commitment to breastfeeding; 3) provide parent education about the infant regarding breastfeeding; 4) provide/find social support needed for continued breastfeeding; and 5) foster linkages to community services that will facilitate the maintenance of breastfeeding.
  The specific activities of the CHN/peer counselor team included hospital visitation after enrollment, home visiting during the first postpartum month, and telephone support throughout the first six postpartum months.
  Arms: 2

SUMMARY:
This research was done to better understand how new mothers who are breastfeeding feel and the questions they have. We wanted to use ways to help new mothers to breastfeed successfully. We compared a new approach (home visits and telephone calls) to the usual care given at Johns Hopkins Hospital with strong support to new mothers from nurses, and a peer counselor (another mother with breastfeeding experience).

DETAILED DESCRIPTION:
Healthy People 2010 included the goal of increasing breastfeeding duration to 6 months for 50% of all mothers. Other professional and national health organizations and the Health and Human Services Blueprint for Action on Breastfeeding recommend that women breastfeed exclusively for six months. Increasing breastfeeding among low-income women is a priority, as disparities exist. Only 20.1% of low-income women (on WIC) breastfeed for six months compared to 40.7 % of more affluent women. Consistent, comprehensive, culturally sensitive breastfeeding support increases duration of breastfeeding, thus offering well-documented health benefits often specifically appropriate for low-income women. Breastfeeding relates to lower formula cost, lower health care costs, and breastfeeding may be less time consuming. These cost savings can potentially offset costs of breastfeeding promotion. Facilitating breastfeeding among low-income women includes comprehensive and culturally relevant support in the hospital, during the first week postpartum, and periodic support in the mother's home. Nearly 35% of low-income women stop breastfeeding within eight days of delivery. Repeated contact with supportive persons such as peer counselors and nurses, affects the duration and exclusivity of breastfeeding practice after the immediate postpartum period. However, support for low-income women has been neglected and not made available because of generally unsubstantiated claims that it is not cost effective. The breastfeeding intervention used an enhanced traditional community health nurse/peer counselor home visit, which is no longer usual care for contemporary community health nursing practice, along with in-hospital and telephone support. The overall hypothesis was the intervention group will have improved breastfeeding outcomes and will demonstrate a net cost savings over usual care.

The consent form explained the purpose of the study; the actual number of visits and telephone calls (if randomized into the intervention group) and the data collecttion procedures. There were no identified risks for those enrolled in the study. Incentives included $105 if the participant completed each data point.

ELIGIBILITY:
Inclusion Criteria:

* breastfeeding
* low-income (WIC eligible)
* English speaking
* telephone available (includes pager or close family member)
* full-term singleton birth, with no cranio-facial abnormalities
* neonate was admitted to the normal newborn nursery (not the NICU)
* negative drug screen for mother and infant.

Exclusion Criteria:

* inability to meet the above criteria

Ages: 12 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 328 (Actual)
Dates: Start 2003-03; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Breastfeeding Rates | March 2003 - August 2006
Breastfeeding duration | March 2003 - August 2006

SECONDARY OUTCOMES:
Cost Implications of a Nurse/Peer Councelor Program | March 2003 - August 2006
Infant indicies related to cost | March 2003 - August 2006

CONTACTS AND LOCATIONS:
Overall Officials: Linda C Pugh, PhD, RNC, FAAN, Principal Investigator — Johns Hopkins University; York College of Pennsylvania
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Result] Frick KD, Milligan RA, White KM, Serwint JR, Pugh LC. Nurse-supported breastfeeding promotion: a framework for economic evaluation. Nurs Econ. 2005 Jul-Aug;23(4):165-72, 206, 147. PMID 16189981
- [Result] Wilson PR, Pugh LC. Promoting nutrition in breastfeeding women. J Obstet Gynecol Neonatal Nurs. 2005 Jan-Feb;34(1):120-4. doi: 10.1177/0884217504272806. PMID 15673655
- [Result] Milligan, R., Low, G., Spatz, D., Brooks, L., Serwint, J., & Pugh, L.C. (2004). Offering breastfeeding mothers advice on contraception. Contemporary Obstetrics & Gynecology, 49.